CLINICAL TRIAL: NCT04780971
Title: Use of Physiology to Evaluate Procedural Result After PCI CTO
Acronym: ULTRA-CTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isala (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Maarten van Leeuwen, Principial Investigator Isala, Isala
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9346
Record Dates: First submitted 2021-01-06; First posted 2021-03-04 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Percutaneous Coronary Revascularisation; Complex Coronary Lesion
Keywords: percutaneous coronary intervention; chronic total occlusion; intra-coronary physiology; optical coherence tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-PCI intra-coronary physiological and OCT measurements (Other): After angiographically successful CTO PCI, intra-coronary physiologic assessment (RFR, FFR, CFR and IMR) and OCT of the CTO vessel will be performed directly. OCT may als be performed during a staged procedure within 4 ± 2 weeks after the index procedure when clinically indicated.
  Interventions: Diagnostic Test: post-PCI Pd/Pa

INTERVENTIONS:
Diagnostic Test: post-PCI Pd/Pa — After angiographically successful CTO PCI, intra-coronary physiologic assessment (RFR, FFR, CFR and IMR) and subsequent OCT of the CTO vessel will be performed. OCT may also be performed during a staged procedure when clinically indicated.
  Other Names: Post-PCI RFR; Post-PCI CFR; Post-PCI IMR; Post-PCI FFR; Post-PCI OCT

SUMMARY:
ULTRA-CTO is a prospective multicentre non-randomised investigator-initiated trial designed to enrol 200 subjects with an indication for percutaneous coronary intervention (PCI) of chronic total occluded (CTO) coronary artery.

The main objective of the study is to assess the predictive value of post-PCI resting full-cycle ratio (RFR) and fractional flow reserve (FFR) with regard to Fractional flow reserve (SSR) in CTO patients.

DETAILED DESCRIPTION:
ULTRA-CTO is a prospective multicentre non-randomised investigator-initiated trial designed to enrol 200 subjects with an indication for PCI CTO.

The main objective of the study is to evaluate both the value of post-PCI RFR and post-PCI FFR for detecting suboptimal stent result (SSR).

After angiographically successful CTO PCI, intra-coronary physiologic assessment (RFR, FFR, coronary flow reserve (CFR) and index of microcirculatory resistance (IMR)) of the CTO vessel will be performed. Additional OCT will be performed directly or during a staged procedure within 4 ± 2 weeks when indicated (i.e. high contrast use, procedural duration, major dissection or other safety reasons according to the operator).

When intra-coronary physiologic assessment or OCT is not possible at all, the patients will not be included in the study.

When the operator decides to optimize the stent result (post-dilation or additional stenting), based on the OCT and/or physiology, post-PCI RFR and FFR should be repeated. For patients undergoing a clinically indicated FFR of a remaining intermediate stenosis (angiographically 30-90%) in a non-CTO vessel or major side branch of the CTO vessel within 4 weeks after the index procedure, intra-coronary physiologic assessment (RFR, FFR, CFR and IMR) will be repeated in the CTO vessel for exploratory objectives

At 4 ± 2 weeks follow-up, the occurrence of cardiovascular events and clinical classification will be assessed for secondary objectives

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older.
2. Angiographically successful PCI CTO without any remaining lesion at least 30% proximal to the stented segment.
3. Possibility to perform physiologic measurements and OCT of sufficient quality.
4. Patients willing and capable to provide written informed consent.

Exclusion Criteria:

1) Contra-indication for adenosine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The AUC of post-PCI RFR compared to the AUC of post-PCI FFR with regard to SSR. | Index procedure (or staged procedure if indicated).
  The AUC of post-PCI RFR compared to the AUC of post-PCI FFR with regard to SSR.

SECONDARY OUTCOMES:
Seattle Angina Questionnaire (SAQ) score at follow-up | 4± 2 weeks
  Seattle Angina Questionnaire (SAQ) score at follow-up
New York Heart Association (NYHA) classification at follow-up | 4± 2 weeks
  New York Heart Association (NYHA) classification (I, II, III or IV) at follow-up
Canadian Cardiovascular Society (CCS) classification at follow-up | 4± 2 weeks
  Canadian Cardiovascular Society (CCS) classification (I, II, III, IV) at follow-up
Occurrence of the composite endpoint of all-cause mortality, myocardial infarction and any coronary revascularization (MACE) at follow-up | 4± 2 weeks
  Occurrence of the composite endpoint of all-cause mortality, myocardial infarction and any coronary revascularization (MACE) at follow-up
The predictive value of the RFR and FFR gradient across the stented segment with regard to SSR in CTO patients. | Index procedure (or staged procedure if indicated).
  The predictive value of the RFR and FFR gradient across the stented segment with regard to SSR in CTO patients.
The correlation between positive RFR (≤0.89) and positive FFR (≤0.80) with regard to SSR following angiographically satisfactory CTO PCI. | Index procedure (or staged procedure if indicated).
  The correlation between positive RFR (≤0.89) and positive FFR (≤0.80) with regard to SSR following angiographically satisfactory CTO PCI.
The correlation between post-PCI physiology (OCT, RFR, FFR, CFR, IMR) and suboptimal stent result (SSR) with anginal complaints (SAQ score), NYHA and CCS classification and MACE at follow-up | Index procedure (or staged procedure if indicated) until 4± 2 weeks follow-up
  The correlation between post-PCI physiology (OCT, RFR, FFR, CFR, IMR) and suboptimal stent result (SSR) with anginal complaints (SAQ score), NYHA and CCS classification and MACE at follow-up.
The impact on physician-decision making based on OCT and physiology findings | Index procedure (or staged procedure if indicated).
  The impact on physician-decision making based on OCT and physiology findings

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Van Leeuwen, PhD, Principal Investigator — Isala Zwolle
Locations (2):
- Netherlands (2):
  - Radboud UMC, Nijmegen
  - Isala, Zwolle

REFERENCES:
- [Derived] Griffioen AM, Meijers TA, Roolvink V, van der Heijden DJ, Volleberg RHJA, van Wely M, van Royen N, van Geuns RJ, van Leeuwen M. Use of physioLogy to evaluaTe procedural Result After percutaneous coronary intervention of Chronic Total Occlusion (ULTRA-CTO): protocol for a prospective, single-arm, multicentre, exploratory study. BMJ Open. 2025 Nov 27;15(11):e108995. doi: 10.1136/bmjopen-2025-108995. PMID 41309467

DOCUMENTS (1):
  • Study Protocol (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT04780971/Prot_000.pdf